CLINICAL TRIAL: NCT02630082
Title: A Cohort Study in Lima, Peru to Evaluate Feasibility of Measuring Immune Responses & Activation Levels in the Foreskin & Rectosigmoid Mucosa in HIV-negative, Uncircumcised Men Who Have Sex With Men & Who Are at High Risk for HIV Acquisition
Brief Title: Feasibility of Measuring Immune Resp, Activation in Foreskin/Mucosa in HIV-, Uncircumcised High-HIV-risk MSM, Lima Peru
Acronym: HVTN 914
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 11704
Record Dates: First submitted 2015-08-24; First posted 2015-12-15 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: HIV Infections; Acquired Immunodeficiency Syndrome; Lentivirus Infections; Retroviridae Infections; RNA Virus Infections; Virus Diseases; Sexually Transmitted Diseases, Viral; Sexually Transmitted Diseases; Immunologic Deficiency Syndromes; Immune System Diseases; Slow Virus Diseases
Keywords: HIV Preventive Vaccine; HIV Seronegativity; Immune Response, Mucosal
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; Lentivirus Infections; Retroviridae Infections; RNA Virus Infections; Virus Diseases; Sexually Transmitted Diseases, Viral; Sexually Transmitted Diseases; Immunologic Deficiency Syndromes; Immune System Diseases; Slow Virus Diseases | interventions — Circumcision, Male

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Other): Circumcision and flexible sigmoidoscopy
  Interventions: Procedure: Circumcision; Procedure: Flexible sigmoidoscopy

INTERVENTIONS:
Procedure: Circumcision
Procedure: Flexible sigmoidoscopy

SUMMARY:
Rectal and genital sampling in HIV prevention trials permits assessments at the site of HIV entry. Yet the safety and acceptability of circumcision and sigmoidoscopy (and associated abstinence recommendations) are unknown in uncircumcised men who have sex with men (MSM) at high risk of HIV infection. The purpose of this study is to evaluate the feasibility of methods for assessing baseline characteristics of the mucosa of MSM at risk of HIV infection in Lima, Peru.

DETAILED DESCRIPTION:
The worldwide HIV/AIDS epidemic may only be controlled through development and utilization of a safe and effective vaccine that will prevent HIV infection. To fill gaps in the understanding of HIV vaccines, studies of mucosal immunity aim to complement assessments of systemic immunity. Yet it is unclear, and important to understand, how mucosal collections and the kinetics of immune activation they might initiate may impact peripheral blood endpoints in HIV vaccine trials. The HIV Vaccine Trials Network (HVTN) and the National Institute of Allergy and Infectious Diseases (NIAID) are conducting a single-site, exploratory cohort study evaluating the feasibility of sampling mucosa and assessing cellular immune responses in sexually active men who have sex with men, a population in which later-phase HIV vaccine clinical trials are often conducted.

The primary purpose of HVTN 914 is to assess the feasibility of performing safe and tolerable circumcision and rectosigmoid biopsy studies on a study population of 30 healthy, HIV-seronegative, uncircumcised men in Lima, Peru, aged 21 to 30 years, who have sex with men and who are at high risk for acquisition of HIV; to assess institutional capacities to process mucosal samples; and to identify methods of evaluating foreskin and rectosigmoid mucosal immune responses that provide minimal variability for analysis of small sample sizes.

The study is designed to mimic an HIV vaccine study mucosal collection protocol. Participants agree to elective sigmoidoscopy biopsy collections and circumcision, and actively participate in this study for approximately 7 months. The primary analysis will focus on pre- and post-procedure retention, safety laboratory values, sexual satisfaction, HIV risk behaviors, and levels of activation markers associated with vulnerability to HIV infection in samples of peripheral blood mononuclear cells. A total of 11 study visits (including a screening visit) occur at Weeks 0-5, 10, and 26-28. Study procedures include physical exams, blood and urine collection, HIV testing, and questionnaire. Elective rectosigmoid bioscopy is performed at Weeks 2 and 27. Elective circumcision is performed at Week 4. Some blood collected from participants will be stored and used in future research. Risk-reduction counseling will be conducted at all study visits.

ELIGIBILITY:
Inclusion Criteria:

1. Male, age 21 to 30 years, who, in the 6 months prior to screening, experienced 1 or both of the following HIV risk criteria:

   * unprotected anal intercourse with 1 or more male or MTF transgender partner(s); or
   * anal intercourse with 2 or more male or MTF transgender partners. Note: Volunteers who have been in a monogamous relationship with an HIV-seronegative partner for > 6 months are excluded.
2. Ability and willingness to provide informed consent
3. Assessment of understanding: volunteer demonstrates understanding of the procedures and purpose of this study. Participants will complete a questionnaire prior to enrollment with verbal demonstration of understanding of all questionnaire items answered incorrectly.
4. Willingness to receive HIV test results
5. Willingness to discuss HIV infection risks (including sexual behavior and drug use) and amenable to HIV risk reduction counseling
6. Willingness to undergo phlebotomy, rectal swab, sigmoidoscopy, and circumcision
7. Willingness to adhere to safety protocols before and after sigmoidoscopy and circumcision
8. Agrees not to enroll in another study of an investigational research agent prior to completion of the last required protocol clinic visit
9. Hemoglobin ≥ 13.0 g/dL
10. White blood cell (WBC) count = 3300 to 12,000 cells/mm3
11. Total lymphocyte count ≥ 800 cells/mm3
12. Remaining differential either within institutional normal range or with site physician approval
13. Platelets = 125,000 to 550,000/mm3
14. Prothrombin time (PT) or partial thromboplastin time (PTT) ≤ 1.25 institutional upper limit of normal; International Normalized Ratio (INR) ≤ 1.5
15. Negative HIV-1 and -2 blood test: May use locally available assays that have been approved by HVTN Laboratory Operations.

Exclusion Criteria:

1. Volunteers who, in the six months prior to screening, have had sexual partners known to be HIV-infected
2. Volunteers who, for the 6 months prior to screening, have been in a monogamous relationship with an HIV-seronegative partner
3. History of immunodeficiency
4. Foreskin covering less than half the glans
5. Absolute medical indication for circumcision (balanitis or phimosis)
6. Bleeding disorder diagnosed by a doctor (eg, factor deficiency, coagulopathy, or platelet disorder requiring special precautions). [This exclusion also applies to therapeutic anticoagulation that results in a prolonged PT/INR or PTT.]
7. HIV vaccine(s) received in a prior HIV vaccine trial. For potential participants who received control/placebo in an HIV vaccine trial, the HVTN 914 PSRT will determine eligibility on a case-by-case basis
8. Untreated clinical signs or symptoms of genitourinary or colonic infection
9. Any medical condition contraindicating circumcision or flexible sigmoidoscopy with biopsies
10. History of transactional sex (ie, exchange of sex for money, shelter, food, or drugs) in the preceding 6 months
11. Any medical, psychiatric, occupational, or other condition that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety, or a participant's ability to give informed consent
12. History of keloid scarring

Ages: 21 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2011-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Pre- and post-procedure retention | 28 weeks
  Number of enrolled trial participants that underwent each procedure visit and attended each follow-up visit
White blood cell counts | 28 weeks
  White blood cells per mm^3
Hematocrit | 28 weeks
  Hematocrit values measured as percentage
Hemoglobin | 28 weeks
  Hemoglobin g/dL
Sexual satisfaction | 28 weeks
  Sexual satisfaction during receptive, insertive sex, and abstinence periods using a CASI behavioral questionnaire (5 point Likert Scale)
HIV risk behaviors | 28 weeks
  Sex without a condom according to a CASI behavioral questionnaire (Yes, No)
Levels of activation markers associated with vulnerability to HIV infection | 28 weeks
  Levels of CCR5, ki67+ Bcl2low, and integrin alpha4beta7 expression on CD4+ CD3+ T cells collected in blood
Procedure-related events | 28 weeks
  Number of procedure related events such as adverse drug reactions, hermorrage/hematoma, infection, pain, perforation/anatomic injury, and edema assessed for severity (NIH/NIAID DIvision of AIDS table for Grading of Severity of Adult and Pediatric Adverse Experiences).
Number of operational protocol deviations per mucosal sample | through study completion, an average of 7 months
  Number of deviations per mucosal sample
Proportion of mucosal samples that are evaluable | through study completion, an average of 7 months
  Percent of total samples (%)
Inter-person variability in mucosal responses | 28 weeks
  Median and range of variables in peripheral blood mononuclear cells, foreskin, and rectosigmoid mucosa
Intra-person differences in mucosal responses obtained from the rectosigmoid colon | 28 weeks
  Median and range of variables in peripheral blood mononuclear cells, foreskin, and rectosigmoid mucosa
Number of clinical protocol deviations per mucosal sample | through study completion, an average of 7 months
  Number of deviations per mucosal sample
Number of laboratory protocol deviations per mucosal sample | through study completion, an average of 7 months
  Number of deviations per mucosal sample

REFERENCES:
- [Derived] Lama JR, Karuna ST, Grant SP, Swann EM, Ganoza C, Segura P, Montano SM, Lacherre M, De Rosa SC, Buchbinder S, Sanchez J, McElrath MJ, Lemos MP; HVTN 914 Study Team. Transient Peripheral Immune Activation follows Elective Sigmoidoscopy or Circumcision in a Cohort Study of MSM at Risk of HIV Infection. PLoS One. 2016 Aug 18;11(8):e0160487. doi: 10.1371/journal.pone.0160487. eCollection 2016. PMID 27536938